CLINICAL TRIAL: NCT05888610
Title: Identifying Specifications for Caregiver-assisted Solutions to Assess Dementia Patient Needs at Home
Brief Title: Caregiver Solutions for Dementia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prepped Health LLC (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 00109123
Record Dates: First submitted 2023-05-10; First posted 2023-06-05 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer's Disease; Dementia; Caregivers; Remote Monitoring
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Outpost (Experimental)
  Interventions: Behavioral: Digital Outpost

INTERVENTIONS:
Behavioral: Digital Outpost — A mobile application that allows caregivers of patients diagnosed with Alzheimer's Disease and Related Dementias to report patient symptom remotely to their clinical team.

SUMMARY:
The goal of this clinical trial is to test a mobile application amongst caregiver's supporting patients diagnosed with Alzheimer's Disease and Related Dementias (ADRD). The main question it aims to answer is: Will caregivers supporting patients diagnosed with ADRD utilize a mobile application to routinely report symptoms of the patients they care for?

ELIGIBILITY:
Inclusion Criteria:

* Caregiver of a Duke patient with Alzheimer's disease or Alzheimer's disease-related dementias (ADRD), participating in the Duke Dementia Family Support Program
* The ability to speak and understand English
* Age > 18 years

Exclusion Criteria:

* Those unable to speak and understand English
* Age ≤ 18 years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Number of Days that Participants Use Digital Outpost | Time Frame up to week 2
  Completion of at least 75% of Digital Outpost across 4 days within a 2-week period
Number of Clinical Assessments Completed | Time Frame up to week 2
  Completion of at least 75% of Clinical Assessments

SECONDARY OUTCOMES:
Usability as Measured by the System Usability Scale at 2 weeks | Time Frame 2 weeks
  The System Usability Scale will be used for rating technology usability. The measure has 10 items. Each item is measured on a 10-point scale ranging from 0-10. The total score ranges from 0-100, where higher scores indicate greater usability.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States